CLINICAL TRIAL: NCT05450042
Title: Scientific Proposal to Substantiate Vascular Effects Through Sirolimus vs. Paclitaxel DCB Implantation
Brief Title: Vascular Effects Through Sirolimus vs. Paclitaxel DCB Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Chistos Rammos, Prof. Dr. med. C. Rammos, MD, FESC, MHBA, University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The Limus FLOW Study
Record Dates: First submitted 2022-06-02; First posted 2022-07-08 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Peripheral Arterial Disease; Flow-mediated Dilation; Drug Eluting Balloon; Infrainguinal Peripheral Arterial Disease
Keywords: Paclitaxel eluting ballon; Sirolimus eluting ballon; Percutaneous transluminal angioplasty
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SELUTION SLR DCB (Experimental): Sustained Limus Release drug eluting balloon
  Interventions: Device: SELUTION SLR DCB
- Paclitaxel eluting balloon (Active Comparator): Conventional: Medtronic INpact
  Interventions: Device: Paclitaxel DCB

INTERVENTIONS:
Device: SELUTION SLR DCB — Sirolimus DCB
  Arms: SELUTION SLR DCB
Device: Paclitaxel DCB — Paclitaxel DCB
  Arms: Paclitaxel eluting balloon

SUMMARY:
Endovascular treatment of symptomatic atherosclerotic peripheral artery disease (PAD) is recommended as the primary revascularization strategy. Percutaneous transluminal angioplasty (PTA) of the superficial femoral artery has a high initial success rate, but restenosis and dissections frequently occur.The influence of the novel devices with improved hemodynamic capabilities with respect to vasomotion of the vessel wall, vascular function and vascular compliance can be measured by FMD (flow-mediated dilation), arterial stiffness indices and vascular strain analysis. The aim of this ITT is to determine the potential improvement and impact of the SELUTION SLR in the infrainguinal arteries on local vascular function.

DETAILED DESCRIPTION:
Endovascular treatment of symptomatic atherosclerotic peripheral artery disease (PAD) is recommended as the primary revascularization strategy. Percutaneous transluminal angioplasty (PTA) of the superficial femoral artery has a high initial success rate, but restenosis and dissections frequently occur. While restoration of tissue perfusion is achieved, these interventional strategies affect vascular function, perpetuating dysfunctional vascular homeostasis. Vascular and endothelial dysfunction per se is the pathophysiologic principle involved in the initiation and progression of atherosclerosis and has been correlated to higher incidences of cardiac events such as myocardial infarction or the need for interventions. PTA and DCB treatment alter the endothelial homeostasis but the impact and detailed mechanisms are incompletely understood. The influence of the novel devices with improved hemodynamic capabilities with respect to vasomotion of the vessel wall, vascular function and vascular compliance can be measured by FMD (flow-mediated dilation), arterial stiffness indices and vascular strain analysis.

The aim of this ITT is to determine the potential improvement and impact of the SELUTION SLR in the infrainguinal arteries on local vascular function.

Device to be used are SELUTION SLR™ (Sustained Limus Release) drug eluting balloon (n = 35) vs. Active comparator, Paclitaxel eluting balloon (Medtronic InPact, n = 35)

The analysis of the primary end point will be performed on an intention-to-treat basis.

Subgroup analyses will be performed according to PAD classification etiology and based on stent length.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral artery disease
* Target lesions 3 cm distal to the CFA-bifurcation including SFA and PA lesions
* Clinical diagnosis of chronic, symptomatic lower limb ischemia as defined by Rutherford 2, 3, 4 and 5
* Planed peripheral intervention TASC A-D
* Subject must be between 18 and 85 years old
* Female of childbearing potential must have a negative pregnancy test within 10 days prior to index procedure and utilize reliable birth control until completion of the 12-month angiographic evaluation
* Vessel diameter ≥4.0 mm and ≤7.0 mm
* Willing to comply with the specified follow-up evaluation
* Written informed consent prior to any study procedures
* Pretreatment with an adequately sized balloon

Exclusion Criteria:

* Bifurcational lesions of the CFA and lesions including the first 3 cm of the SFA, due to technical aspects of FMD measurement
* Instent-Restenosis
* Thrombolysis within 72 hours prior to the index procedure
* Aneurysm formations in the femoral artery or popliteal artery
* Concomitant hepatic insufficiency, deep venous thrombus, coagulation disorder or receiving immunosuppressant therapy
* Unstable angina pectoris at the time of the enrollment
* Recent myocardial infarction or stroke < 30 days prior to the index procedure
* Life expectancy less than 12 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-04-06 (Estimated); Study Completion 2024-04-06 (Estimated)

PRIMARY OUTCOMES:
Change of flow-mediated vasodilation (FMD) of the nonstenotic segment of the proximal SFA after procedure | 1 month
  FMD represents the percent diameter gain as calculated based on preischemia and postischemia diameter measurements of the femoral artery
Change of flow-mediated vasodilation (FMD) of the nonstenotic segment of the proximal SFA after procedure | 6 months
  FMD represents the percent diameter gain as calculated based on preischemia and postischemia diameter measurements of the femoral artery
Change of flow-mediated vasodilation (FMD) of the nonstenotic segment of the proximal SFA after procedure | 12 months
  FMD represents the percent diameter gain as calculated based on preischemia and postischemia diameter measurements of the femoral artery

SECONDARY OUTCOMES:
Changes in pulse wave velocity (PWV) | Baseline, followed at 1, 6 and 12 months
  Changes in cardiovascular function measured by pulse wave velocity in m/s
Changes in augmentation index | Baseline, followed at 1, 6 and 12 months
  Changes in cardiovascular function measured by augmentation index in %
Changes in vascular strain | Baseline, followed at 1, 6 and 12 months
  Changes in cardiovascular function measured by vascular strain in %
Changes in peripheral perfusion determined by ABI (ankle brachial index) | Baseline, followed at 1, 6 and 12 months
  ABI measurements are conducted using a Doppler probe on tibial and anterior artery locations. The highest value will be used for calculation and divided by the highest systolic brachial Doppler pressure
Primary patency (PP) of target lesion | Baseline, followed at 1, 6 and 12 months
  Primary patency determined by PVR measurement with ultrasound
Changes in clinical symptoms | Baseline, followed at 1, 6 and 12 months
  Clinical symptoms of patients determined by Walking impairment questionaire (WIQ)
Changes in six-minute walk test | Baseline, followed at 1, 6 and 12 months
  Six-minute walk test determined by pain-free walking distance in m
Procedural complications | Baseline, followed at 1, 6 and 12 months
  Any procedural complications
Freedom from Target Lesion Revascularization | Baseline, followed at 1, 6 and 12 months
  Freedom from Target Lesion Revascularization (FTLR)
MALE | Baseline, followed at 1, 6 and 12 months
  Any unplanned vascular event and minor or major amputations
Changes of inflammatory profile measured by hs-CRP in mg/dl | Baseline, followed at 1, 6 and 12 months
  Blood samples are collected at the below mentioned time points
Changes of inflammatory profile measured by oxLDL in µg/l | Baseline, followed at 1, 6 and 12 months
  Blood samples are collected at the below mentioned time points
Changes of inflammatory profile measured by Interleukin-6 in pg/ml | Baseline, followed at 1, 6 and 12 months
  Blood samples are collected at the below mentioned time points

CONTACTS AND LOCATIONS:
Overall Officials: Christos Rammos, Professor, Principal Investigator — University Hospital, Essen
Locations (1):
- University of Essen, Clinic of Cardiology and Angiology, Essen, North Rhine-Westphalia, Germany